CLINICAL TRIAL: NCT02218099
Title: A Phase 1 Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics, Pharmacodynamics and Safety of ASP8232 (Part 1) and a Multiple Dose, Placebo-controlled Exploratory Safety, Pharmacokinetic and Pharmacodynamic Study in Type 2 Diabetes Mellitus Subjects With Chronic Kidney Disease (Part 2)
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of ASP8232 in Subjects With Renal Impairment and in Type 2 Diabetes Mellitus Subjects With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 8232-CL-0002; 2013-000680-89 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP8232; Pharmacodynamics of ASP8232; Chronic Kidney Disease (CKD); Type 2 Diabetes Mellitus (T2DM)
Keywords: ASP8232; Multiple doses; Phase 1; Single dose
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — ASP8232

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Single dose of ASP8232 (Experimental): Subjects receive a single oral dose of ASP8232
  Interventions: Drug: ASP8232
- 2: Multiple doses of ASP8232 or placebo (Experimental): Subjects receive multiple oral doses of ASP8232 or placebo
  Interventions: Drug: ASP8232; Drug: Placebo

INTERVENTIONS:
Drug: ASP8232 — Oral
Drug: Placebo — Oral
  Arms: 2: Multiple doses of ASP8232 or placebo

SUMMARY:
This study consists of two parts.

Part 1 evaluates the effect of renal impairment on the PK and PD of a single dose of ASP8232. In addition, the safety and tolerability will be assessed.

Part 2 evaluates the PK, PD, and safety and tolerability of multiple doses of ASP8232 compared with placebo in Type 2 Diabetes Mellitus (T2DM) subjects with Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
This is a two-part study. Part 1 compares the pharmacokinetics (PK), pharmacodynamics (PD) and safety and tolerability of ASP8232 in healthy subjects with subjects with different degrees of renal impairment; Part 2 is a multiple-dose, placebo-controlled study to evaluate the PK, PD and safety and tolerability of multiple doses of ASP8232 in T2DM subjects with CKD.

Part 1:

Subjects reside in the clinic for 9 days, receiving a single oral dose of ASP8232 on Day 1 under fasted conditions followed by a 168-hours blood and urine PK/PD sampling period. Subjects are discharged on Day 8 and return to the clinic on Days 10, 12, 14, 21, 28, and 42 for the collection of blood PK/PD samples. An End of Study Visit (ESV) takes place after the last PK sample is collected on Day 56.

Part 2:

Subjects are admitted to the clinic on Day -2 in order to collect PD urine samples before dosing begins on Day 1. Subjects receive multiple oral doses of ASP8232 or placebo for 28 days. They are discharged on Day 8 and return to the clinic on Days 14 and 21, and Days 27 to 29 for blood PK/PD and urine PD samples. An ESV takes place 14 to 28 days after the last PK/PD sample is collected.

ELIGIBILITY:
Main Inclusion: Part 1

* Independent Ethics Committee (IEC)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the study period and for 28 days (or 5 half-lives of the study drug whichever is longer) after final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for at least 90 days after final study drug administration.
* Female subject must be either:

  * post-menopausal (defined as at least one year without any menses) prior to screening, or
  * premenarchal prior to screening, or
  * documented surgically sterile or status post hysterectomy (at least 1 month before screening), or
  * if of childbearing potential, must have a negative urine pregnancy test at screening and must be using highly effective contraception. All females of childbearing potential will be required to use highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and throughout the study period and for 28 days (or 5 half-lives of the study drug whichever is longer) after final study drug administration.
* Female subject must not be lactating, and must not be breast feeding at screening or during the study period and for 28 days [or 5 half-lives of the study drug whichever is longer] after final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days [or 5 half-lives of the study drug whichever is longer] after final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Healthy Subjects:

* Subject must have pre dose eGFR values (based on the MDRD method) at screening and day -1 higher or equal to 80 mL/min/1.73 m2.

Renal Impaired Subjects:

* Subject must have pre dose eGFR values (based on the MDRD method) at screening and day -1 of 15 to < 30 mL/min/1.73 m2, 30 to

< 60 mL/min/1.73 m2 or 60 to < 80 mL/min/1.73 m2 for severe, moderate or mild renal impaired subjects, respectively.

Part 2 Inclusion:

* Independent Ethics Committee (IEC)-approved written Informed Consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
* Subject has either known or confirmed T2DM with CKD for at least 1 year [screening].
* Subject is ≥ 35 and ≤ 80 years of age.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continue throughout the study period and for 28 days (or 5 half-lives of the study drug whichever is longer) after final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for at least 90 days after final study drug administration.
* Female subject must be either

  * post-menopausal (defined as at least one year without any menses) prior to Screening, or
  * premenarchal prior to screening, or
  * documented surgically sterile or status post hysterectomy (at least 1 month before screening), or
  * if of childbearing potential, must have a negative urine pregnancy test at screening and must be using highly effective contraception1. All females of childbearing potential will be required to use highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and throughout the study period and for 28 days (or 5 half-lives of the study drug whichever is longer) after final study drug administration.
* Female subject must not be lactating, and must not be breast feeding at screening or during the study period and for 28 days (or 5 half-lives of the study drug whichever is longer) after final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 28 days (or 5 half-lives of the study drug whichever is longer] after final study drug administration.
* Subject is on a stable therapy with ACE inhibitors or ARB for at least 3 months [screening].
* Subject is on a stable anti-hyperglycaemia therapy, e.g. with Metformin, SUD, TZD or DPP-4 inhibitor.
* Subject's eGFR is between 15-60 mL/min/1.73 m2 (based on the MDRD method).
* Subject's HbA1c level is lower than 7.5% at clinic admission on day -2.
* Subject has a stable blood pressure for at least 3 to 6 months prior to enrolment.
* Subject's UACR is higher than 30 mg/g at clinic admission on day -2.

Part 1 Exclusion:

All Subjects:

* Female subject who has been pregnant within 6 months before screening or breast feeding within 3 months before screening.
* Subject has a known or suspected hypersensitivity to ASP8232, or any components of the formulation used.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has Gilbert's syndrome.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check in.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14 units of alcohol for female subjects) within 3 months prior to admission to the Clinical Unit.
* Subject uses drugs of abuse within 3 months prior to admission to the Clinical Unit.
* Subject regularly uses any inducer of metabolism (e.g. barbiturates, rifampin ) in the 3 months prior to admission to the Clinical Unit.
* Subject had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on day -1.
* Subject has positive serology test for Hepatitis B Surface Antigen (HBsAg), anti-Hepatitis A virus (anti-HAV [IgM]), anti-Hepatitis C virus (anti-HCV) or anti- Human immunodeficiency virus 1 + 2 (anti-HIV 1+2).
* Subject participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives whichever is longer, prior to the initiation of screening.
* Subject is an employee of the Astellas Group or Clinical Research Organization (CRO) involved in the study.

Healthy Subjects:

* Subject has any of the liver function tests (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], total bilirubin [TBL]) above the upper limit of normal. In such a case the assessment may be repeated once [day -1].
* Subject has a mean QTc(F) interval of > 430 ms (for males) and > 450 ms (for females) at screening and day -1. If the mean QTc(F) exceeds the limits above, one additional triplicate electrocardiogram (ECG) can be taken. If this triplicate also gives abnormal result the subject should be excluded.
* Subject uses any prescribed or non-prescribed drugs (including vitamins, hormone replacement therapy, natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day).

Renal Impaired Subjects:

* Subject is on or requires hemodialysis or has received a kidney transplantation.
* Subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 100 mmHg, or pulse rate < 40 or > 90 beats p/m, on screening and day -1. In such a case the assessment may be repeated once (day -1).
* Subject has a mean QTc(F) interval of > 450 ms (for males) and > 470 ms (for females) at screening and day -1. If the mean QTc(F) exceeds the limits above, one additional triplicate ECG can be taken. If this triplicate also gives abnormal result the subject should be excluded.
* Subject has not been on a stable dose of allowed concomitant medications for at least 2 weeks prior to day 1 and/or for whom dose changes are likely to occur during the study.
* Subject requires or is likely to require any new concomitant medications during the course of the study.
* Subject has obstructive uropathy or other causes of renal impairment not related to parenchymal renal disorder and/or disease of the kidney.
* Subject has renal disease secondary to malignancy.
* Subject has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to screening, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the screening period.
* Subject has any of the liver function tests (ALT, AST, TBL) out of range. In such a case the assessment may be repeated once [day -1].

  * ALT or AST > 2 x upper limit of normal (ULN)
  * TBL > 1.5 x ULN

Part 2 Exclusion

* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has known or suspected hypersensitivity to ASP8232 or sinistrin, or any components of the formulation used.
* Subject has participated in part 1 of the 8232-CL-0002 study.
* Subject has a mean QTc(F) interval of > 450 ms (for males) and > 470 ms (for females) at screening and day -2. If the mean QTc(F) exceeds the limits above, one additional triplicate ECG can be taken. If this triplicate also gives abnormal result the subject should be excluded.
* Subject has a pulse < 40 or > 90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically) at screening and day -2. In such a case the assessment may be repeated once [day -2].
* Subject is on or requires hemodialysis or has received a kidney transplantation.
* Subject has not been on a stable dose of allowed concomitant medications for at least 2 weeks prior to day 1 and/or for whom dose changes are likely to occur during the study.
* Subject who requires or is likely to require any new concomitant medications during the course of the study.
* Subject who has obstructive uropathy or other causes of renal impairment not related to parenchymal renal disorder and/or disease of the kidney.
* Subject who has renal disease secondary to malignancy.
* Subject who has a fluctuating or rapidly deteriorating renal function within 4 weeks prior to the study, as indicated by strongly varying or worsening of clinical and/or laboratory signs of renal impairment within the screening period.
* Subject has type 1 diabetes mellitus.
* Subject with any of the liver function tests (ALT, AST, TBL) out of range as indicated below. In such a case the assessment may be repeated once [day -2].

  * ALT or AST > 2 x ULN
  * Total bilirubin > 1.5 x ULN
* Subject has had myocardial infarct or stroke within 6 months prior to screening.
* The subject has Gilbert's Syndrome.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within one week prior to clinic admission on day -2.
* Subject has a history of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14 units of alcohol for female subjects) within 3 months prior to admission to the Clinical Unit.
* Subject uses of drugs of abuse within 3 months prior to admission to the Clinical Unit.
* Subject regularly uses any inducer of metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
* Subject had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on day -2.
* Subject has positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.
* Subject participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives whichever is longer, prior to the initiation of screening.
* Subject is employee of the Astellas Group or CRO involved in the study.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
Part 1: PK of ASP8232 in plasma measured by Area Under the concentration-time Curve (AUC) from zero to infinity with extrapolation of the terminal phase (AUCinf) | Day 1 to Day 56
Part 1: PK of ASP8232 in plasma measured by AUC from zero up to last time point of observation (AUClast) | Day 1 to Day 56
Part 1: PK of ASP8232 in plasma measured by AUC from zero up to last time point of observation, unbound fraction (AUClast,u) | Day 1 to Day 56
Part 1: PK of ASP8232 in plasma measured by AUC from 0 to infinity with extrapolation of the terminal phase, unbound fraction (AUCinf,u) | Day 1 to Day 56
Part 1: PK of ASP8232 in plasma measured by maximum concentration (Cmax) | Day 1 to Day 56
Part 1: PK of ASP8232 in plasma measured by maximum concentration, unbound fraction (Cmax,u) | Day 1 to Day 56
Part 2: Safety and tolerability of ASP8232 measured by nature, frequency and severity of AEs, vital signs, safety laboratory tests, routine ECG | Screening to End of Study Visit (ESV)

SECONDARY OUTCOMES:
Part 1: PK profile of ASP8232 in plasma | Day 1 to Day 56
  apparent total plasma clearance of drug after oral administration (CL/F), renal clearance based on unbound plasma concentrations (CLu/F), fraction unbound (fu), lag-time (time delay between drug administration and first observed concentration above LOQ in plasma) (tlag), time to reach Cmax (tmax), terminal elimination half-life (t1/2), apparent volume of distribution during terminal phase after oral administration (Vz/F), apparent volume of distribution during terminal phase after oral administration, unbound fraction (Vz,u/F)
Part 1: PK profile of ASP8232 in urine | Day -1 to Day 8
  renal clearance (CLR), CLR unbound fraction (CLR,u), amount of drug excreted in urine from time point 0 to time point 24 h (Ae0-24h), percent of drug excreted in urine from time point 0 to time point 24 h (Ae0-24h%), cumulative amount of drug excreted in urine from time of dosing up to the collection time of the last measurable concentration (Aelast), percent of drug dose excreted in urine (Aelast) from time of dosing up to the collection time of the last measurable concentration (Aelast%), cumulative amount of drug excreted in urine from time of dosing extrapolated to time infinity (Aeinf), percent of drug dose excreted in urine (Aeinf) from time of dosing extrapolated to time infinity (Aeinf%)
Part 1: PD of Vascular adhesion protein-1 (VAP-1) activity in plasma | Day -1 to Day 56
  maximum activity (Rmax), maximum activity in percent (Rmax%), time to attain maximal Response (tmax, R), average response over the first 24 h after dosing (Ravg, 0-24h)
Part 1: PD of Total antioxidant status (TAS) in serum | Day -1 to Day 56
  Rmax, Rmax%, tmax, R, Ravg, 0-24h
Part 1: Safety and tolerability of ASP8232 | Screening to Day 56
  nature, frequency and severity of Adverse Events (AEs), vital signs, safety laboratory tests, routine Electrocardiogram (ECG)
Part 2: PK profile of ASP8232 in plasma | Day 1 to Day 29
  free drug fraction (fu), area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau), area under the concentration-time curve during a dosing interval at steady state, unbound fraction (AUCtau,u), tmax, Cmax, Cmax,u, CL/F, CLu/F, Peak Trough Ratio (PTR), concentration immediately prior to dosing at multiple dosing (Ctrough), Ctrough, unbound (Ctrough, u)
Part 2: PK profile of ASP8232 in urine | Day 1 to Day 8 and Day 28 to Day 29
  amount of unchanged drug excreted in urine over a dosing interval in steady state (Aetau), amount of unchanged drug excreted in urine over a dosing interval in steady state in % (Aetau%), CLR, CLR,u
Part 2: PD of VAP-1 activity in plasma | Day -2 to Day 21 and Day 28 to ESV
  Rmax and Rmax%
Part 2: PD of TAS in serum | Day -2 to Day 21 and Day 28 to ESV
  Rmax, Rmax%, tmax, R, Ravg, 0-24h
Part 2: 24-hour urinary albumin excretion rate (UAER) | Day -1, Day 7 and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Central contact, Study Director — Astellas Pharma Europe B.V.
Locations (3):
- Site: 35901, Sofia, Bulgaria
- Site: 37301, Chisinau, Moldova
- Site: 40001, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=314